CLINICAL TRIAL: NCT05287919
Title: Effects of Low- and Medium-frequency Neuromuscular Electrical Stimulation on Skeletal Muscle Atrophy in Critically Ill Patients
Brief Title: Neuromuscular Electrical Stimulation (NMES) Preserves Muscle Mass in Intensive Care Unit (ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabriel Nasri Marzuca-Nassr (Other)
Responsible Party: Sponsor-Investigator, Gabriel Nasri Marzuca-Nassr, Professor, Universidad de La Frontera
Organization: Universidad de La Frontera (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tesis UFRO #1676
Record Dates: First submitted 2022-02-19; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness; Physical Disability; Muscle Atrophy
Keywords: electrical stimulation therapy; skeletal muscle atrophy; critically ill patient; physical therapy; intensive care unit
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Patients received the standard physical therapy (SPT) programme only (passive mobilization) twice a day.
  Interventions: Other: Patients received the standard physical therapy (SPT) programme (passive mobilization) twice a day.
- Low-frequency NMES group (Experimental): Patients submitted to low-frequency NMES and SPT twice a day.
  Interventions: Other: Patients received the standard physical therapy (SPT) programme (passive mobilization) twice a day.; Other: Patients received the low-frequency neuromuscular electrical stimulation (NMES)
- Medium-frequency NMES group (Experimental): Patients submitted to medium-frequency NMES and SPT twice a day.
  Interventions: Other: Patients received the standard physical therapy (SPT) programme (passive mobilization) twice a day.; Other: Patients received the medium-frequency neuromuscular electrical stimulation (NMES)

INTERVENTIONS:
Other: Patients received the standard physical therapy (SPT) programme (passive mobilization) twice a day. — All participants have received standard physical therapy (SPT) sessions based on a passive range of motion mobilization protocol for the lower limbs. It consisted of a bilateral series of 10 repetitions of hip flexion, knee flexion and extension, and ankle flexion and extension. The procedure was performed twice a day: a morning (between 8am - 12pm) and an afternoon session (between 2pm - 6pm).
Other: Patients received the low-frequency neuromuscular electrical stimulation (NMES) — Electrical stimulation was performed twice a day after SPT. Two electrodes were attached to each thigh at the motor points of the quadriceps muscle. The point halfway between the anterior superior iliac spine and the base of the patella was used as reference and electrodes were placed 15 cm apart each other, 5 cm proximal and 10 cm distal from the reference point. After the first measurement, semi-permanent markers were used to indicate the position of electrodes. Electrical stimulation was performed using a 4-channels device (Sonopuls 492, series 4, Enraf-Nonius®, Rotterdam, Netherlands). The low-frequency protocol consisted of 100 Hz and 400 ms width pulses, delivered in trains of 5 s ON (ramp-up time: 1 s, plateau: 3 s, ramp-down time: 1 s) and 10 s OFF. Sessions had 20 min of duration (total of 40 min/day) and the current amplitude (mA) was adjusted to the identification of visible and palpable contractions and was rectified every 3 min to sustain the initial level of contraction.
  Arms: Low-frequency NMES group
Other: Patients received the medium-frequency neuromuscular electrical stimulation (NMES) — Electrical stimulation was performed twice a day after SPT. Two electrodes were attached to each thigh at the motor points of the quadriceps muscle. The point halfway between the anterior superior iliac spine and the base of the patella was used as reference and electrodes were placed 15 cm apart each other, 5 cm proximal and 10 cm distal from the reference point. After the first measurement, semi-permanent markers were used to indicate the position of electrodes. Electrical stimulation was performed using a 4-channels device (Sonopuls 492, series 4, Enraf-Nonius®, Rotterdam, Netherlands).The medium-frequency protocol had similar parameters, but a carrier frequency of 2500 Hz and burst frequency of 100 Hz. Sessions had 20 min of duration (total of 40 min/day) and the current amplitude (mA) was adjusted to the identification of visible and palpable contractions and was rectified every 3 min to sustain the initial level of contraction.
  Arms: Medium-frequency NMES group

SUMMARY:
Background: Low-frequency neuromuscular electrical stimulation (NMES) attenuates the loss of muscle mass of Intensive Care Unit (ICU) patients. However, it has been shown that medium-frequency NMES may be better than low-frequency for the maintenance of skeletal muscle mass in healthy subjects.

Objective: to compare the effects of low-frequency and medium-frequency NMES, along with a standard physical therapy (SPT) programme, on the attenuation of skeletal muscle atrophy in critically ill patients.

Methods: Fifty-four critically ill patients admitted into intensive care unit (ICU) and on mechanical ventilation (MV) participated in this randomized, single-blinded, experimental study. Participants were allocated to one of the following groups: Control Group (CG), received a standard lower limb physical therapy (SPT) programme, 2x/day; Low-frequency NMES Group (LFG), received lower limb SPT+NMES at 100 Hz, 2x/day; and Medium-frequency NMES Group (MFG), received lower limb SPT+NMES at 100 Hz and carrier frequency of 2500 Hz, 2x/day. The primary outcome was the thickness and quality of the quadriceps muscle, evaluated with ultrasonography while patients were in ICU. Secondary outcomes, assessed at various stages of recovery, were strength, functionality, independence for activities of daily living, quality of life, and total days hospitalized.

DETAILED DESCRIPTION:
Background: Low-frequency neuromuscular electrical stimulation (NMES) attenuates the loss of muscle mass of Intensive Care Unit (ICU) patients. However, it has been shown that medium-frequency NMES may be better than low-frequency for the maintenance of skeletal muscle mass in healthy subjects.

Research question: The research question was is medium-frequency neuromuscular electrical stimulation (NMES) more effective than low-frequency NMES for the attenuation of skeletal muscle atrophy in critically ill patients?

Objective: To compare the effects of low-frequency and medium-frequency NMES, along with a standard physical therapy (SPT) programme, on the attenuation of skeletal muscle atrophy in critically ill patients.

Methods: Fifty-four critically ill patients admitted into intensive care unit (ICU) and on mechanical ventilation (MV) participated in this randomized, single-blinded, experimental study. Participants were allocated to one of the following groups: Control Group (CG), received a standard lower limb physical therapy (SPT) programme, 2x/day; Low-frequency NMES Group (LFG), received lower limb SPT+NMES at 100 Hz, 2x/day; and Medium-frequency NMES Group (MFG), received lower limb SPT+NMES at 100 Hz and carrier frequency of 2500 Hz, 2x/day. The primary outcome was the thickness and quality of the quadriceps muscle, evaluated with ultrasonography while patients were in ICU. Secondary outcomes, assessed at various stages of recovery, were muscle strength (MRC-SS), handgrip strength (dynamometry), functional status (FSS-ICU), degree of independence for activities of daily living (Barthel Index), functional mobility and dynamic balance (Timed Up and Go Test), quality of life (SF-36), and total days hospitalized.

ELIGIBILITY:
Inclusion Criteria:

- patients between 18-80 years old admitted in ICU with requirement of mechanical ventilation (MV) for longer than 72 h.

Exclusion Criteria:

* non-sedated patients;
* spinal cord injury;
* cerebrovascular accident;
* patients with pacemakers;
* history of deep vein thrombosis;
* pregnancy;
* cardiac complications (history of myocardial infarction or congenital diseases);
* use of neuromuscular blockers;
* polytraumatized patients requiring tutor support.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in thickness of the quadriceps muscle, evaluated with ultrasonography while patients were in intensive critical unit (ICU). | Day 1, Day 5, Day 9
  Thickness of the quadriceps muscle via ultrasonography (mm).
Change in quality of the quadriceps muscle, evaluated with ultrasonography while patients were in intensive critical unit (ICU). | Day 1, Day 5, Day 9
  Quality of the quadriceps muscle via ultrasonography by Heckmatt's rating scale.
  Muscle quality was estimated by Heckmatt's rating scale, which scores the ultrasound images between 1-4: 1) normal echogenicity; 2) slight increase in muscle echogenicity and normal bone reflection; 3) moderate increase in muscle echogenicity and reduced bone reflection; 4) large increase in muscle echogenicity and no bone reflection.

SECONDARY OUTCOMES:
Change in Clinical assessment of muscle strength while patients were in intensive care unit (ICU). | Day 9, Day 11, Day 16, and Day 27
  Clinical assessment of muscle strength via Medical Research Council-Sum Score (MRC-SS) (points), which ranges from 0 (complete paralysis) to 60 (normal strength).
Change in Handgrip strength while patients were in hospital stay. | Day 9, Day 11, Day 16, and Day 27
  Handgrip strength via digital dynamometer (kg).
Change in Functional status while patients were in Intensive Care unit (ICU). | Day 9, Day 11, Day 16, and Day 27
  Functional status via Functional Status Score for the Intensive Care Unit (FSS-ICU) (points). FSS-]ICU FSS-ICU score has a range of 0-35 with higher score indicating better functional status.
Change in dynamic balance while patients were in hospital stay. | Day 16, and Day 27
  Dynamic balance via Timed Up and Go Test (seconds).
Change in independence for activities of daily living while patients were in hospital stay. | Day 16, and Day 27
  Independence for activities of daily living via Barthel index (points). A patient scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities.
Change in quality of life prior to hospital discharge. | Day 27
  Quality of life via Short Form 36 (SF-36) (points). The score go from 0 to 100. Higher scores mean a better outcome.

OTHER OUTCOMES:
Change in days spent in Mechanical Ventilation. | Through mechanical ventilation use completion, an average of 9 days
  Number of days spent in Mechanical Ventilation use.
Change in days spent in Intensive Care Unit. | Through Intensive Care Unit stay completion, an average of 11 days
  Number of days spent in Intensive Care Unit stay.
Change in days spent in the hospital. | Through hospital stay completion, an average of 27 days
  Number of days spent in hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel N Marzuca-Nassr,, PT, MSc, PhD, Principal Investigator — Universidad de La Frontera
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, Universidad de La Frontera, Temuco, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guerra-Vega P, Guzman R, Betancourt C, Grage M, Vera C, Artigas-Arias M, Munoz-Cofre R, Vitzel KF, Marzuca-Nassr GN. Medium-Frequency Neuromuscular Electrical Stimulation in Critically Ill Patients Promoted Larger Functional Capacity Improvement During Recovery than Low-Frequency Neuromuscular Electrical Stimulation: Randomized Clinical Trial. J Clin Med. 2025 Jul 31;14(15):5407. doi: 10.3390/jcm14155407. PMID 40807029